CLINICAL TRIAL: NCT04509830
Title: Efficacy of Hip Strengthening on Dynamic Knee Stability, Disability and Gait in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HebaAllah Elsayed Mohamed Elsaeed, head of physiotherapy department at Benha fever hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hip strength on KOA
Record Dates: First submitted 2020-08-03; First posted 2020-08-12 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hip strengthening (Experimental): resistance training for hip abductor, hip extensor, and hip external rotator will be performed.cuff weights will be used with 80% of 1 repetition maximum at 3 sets of 8 repetitions with 10-15 second rest between repetitions and 1-2 minute rest between sets.
  Interventions: Other: hip strengthening; Other: quadriceps strengthening, stretch hamstring,cuff muscles
- quadriceps strengthening, stretch for hamstring,cuff muscles (Active Comparator): quadriceps strengthening: multi-angle isometric exercise from sitting position will be performed. cuff weights will be used with 3 sets of 12 repetitions at 40% of 1 reprtition maximum.
  self stretch for hamstring and cuff muscles from supine position. the procedure will be repeated 4 times.
  Interventions: Other: quadriceps strengthening, stretch hamstring,cuff muscles

INTERVENTIONS:
Other: hip strengthening — resistance training for hip abductor, hip extensor, and hip external rotator
  Arms: hip strengthening
Other: quadriceps strengthening, stretch hamstring,cuff muscles — multi-angle isometric quadriceps strengthening and hamstring and cuff self stretch

SUMMARY:
this study will be conducted to investigate the role of hip strengthening in improving dynamic knee stability, gait parameter, lower extremity strength and disability in knee osteoarthritis

DETAILED DESCRIPTION:
knee osteoarthritis accounts for more than 80% of the total burden of the diseases. patients with knee osteoarthritis had worse spatiotemporal gait parameter and dynamic instabitity. there are significant hip muscle weakness in knee osteoarthritis. hip muscle weakness leads to improper alignment and stress in knee joint. hip muscle strength can affect knee joint loading and disease progression in knee osteoarthritis. muscles of the lower extremity play a critical role in the preservation of normal knee joint function by providing dynamic knee joint stability and shock absorption, while maintaining safe transfer of forces across the joint.

ELIGIBILITY:
Inclusion Criteria:

age 40 to 65 years grade 2-3 on KL grade BMI 25 to 32 kg/m2 medial KOA

Exclusion Criteria:

* lateral KOA intraarticular corticosteriod injection into knee within pervious 3 months significant comorbidity individuals with known hip osteoarthritis previous trauma affection one or both hips history of other medical conditions affecting the knee joint previous replacement of any joint in the lower extremity low back pain cognitive impairment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
dynamic knee stability | baseline
  dynamic knee stability will be measured by frontal plane projection angle